CLINICAL TRIAL: NCT06442033
Title: Genetics and Aerobic Exercise to Slow Parkinson's Disease (GEARS) Trial
Brief Title: Genetics and Aerobic Exercise to Slow Parkinson's Disease Trial
Acronym: GEARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jay Alberts (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Jay Alberts, Center Director, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-100
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Group
Masking Description: A historical control group will be utilized for analysis from a previous project. All participants in this study will be exercising in the community setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): All participants will exercise in a community setting 3x/week for 12 months
  Interventions: Other: High intensity stationary cycling

INTERVENTIONS:
Other: High intensity stationary cycling — All community based exercise sessions are: 3x/week for 40 min, which includes a 5-min warm up & cool down and a 30-minute main exercise set. Exercise parameters will be set by a neurologically trained physical therapist and will be progressed over time with the ultimate goal of the individual reaching moderate-vigorous exercise. Moderate-vigorous exercise for this project is defined as a cadence of 75+ rpms and a target HR of 60-80% of their age-predicted max

SUMMARY:
The proposed multi-site, Genetics and Aerobic Exercise to Slow PD (GEARS) Trial will, for the first time, determine the interplay between genetics and exercise in altering PD progression. In sum, 200 PD patients will be recruited from the Cleveland and Salt Lake City metro areas to participate in the Pedaling for Parkinson's (PFP) community-based exercise program. Participants will exercise at community-based sites 3x/week for 12 months. All participants will undergo genotyping using an array that includes the genome backbone and common risk variants associated to increase risk for multiple neurological disorders including PD.

DETAILED DESCRIPTION:
A long-standing unmet need in the treatment of Parkinson's disease (PD) is the identification of a disease-modifying intervention (e.g. pharmaceutical, surgical or behavioral). A growing body of evidence indicates that high-intensity aerobic exercise, when delivered in a highly supervised, well-controlled laboratory setting, improves PD symptomology. Two fundamental gaps remain related to the widespread utilization of exercise to slow PD: 1) are community-based exercise programs effective in altering disease progression and 2) what is the role of genetics in modulating the disease altering effects of high-intensity aerobic exercise? Our underlying hypothesis is that high-intensity, community-based exercise slows disease progression in PD and does so more effectively in individuals with a lower genetic/biological burden. Genetic burden for PD will be determined through the calculation of a PD polygenic risk score (PRS).

Total study duration is ~12.5 months to accommodate data collection sessions and enrollment in PFP class. The study consists of five in-person assessments at the Cleveland Clinic or the University of Utah: informed consent, enrollment (On- and Off-medication separated by at least 24 hrs), 6 months (Off-medication), and 12 months (Off-medication). Asking participants to withhold medication for Off-state examinations imposes a burden, but the Off-state (12 hours off meds) will increase insight into the direct effect of exercise on PD and provides more reliable, less confounded time comparisons. Antiparkinsonian medication will be reconciled at Baseline, 6- and 12-month timepoints. Outcome metrics are provided in Table 1. Notably, all outcome metrics will be collected at each time point after the consent appointment (baseline on, baseline off, 6 month and 12 month) with the exception of the quality of life metrics (Neuro-QoL and MDS-UPDRS I, II, IV) which will be collected at one of the two baseline assessments (instead of both baseline assessments), 6 month, and 12 month; the quality of life questionnaires ask questions about one's quality of life over the previous 7 days and are non-specific to medication state. Genetic data and demographics will be gathered at the first enrollment assessment visit. Following the two enrollment visits, the participant will begin attending PFP classes 3x/wk at the community center most convenient to them. Participants will be recruited and enrolled on a continuous basis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult with a diagnosis of PD by a physician or physician extender
2. Hoehn and Yahr stage I-III
3. Demonstrate the ability to safely mount and dismount a stationary cycle
4. Reliable transportation to the community exercise facility
5. Smartphone device for activity data monitoring
6. On a stable dose of anti-parkinsonian medication

Exclusion Criteria:

1. Participation in disease modifying PD-related clinical trial or study
2. Diagnosis of dementia or any neurocognitive impairment that compromises one's ability to provide informed consent.
3. Implanted deep brain stimulation electrodes or focused ultrasound for PD management
4. Recommendation for medical clearance using the American College of Sports Medicine (ACSM) Preparticipation Health Screen a. If the ACSM screen recommends medical clearance, the participant must obtain medical clearance by their health care provider prior to participation.

b. Those who choose not to obtain physician clearance will not be eligible for participation.

e) A musculoskeletal issue (arthritis, osteoporosis, back problem) that would limit one's ability to engage in a cycling intervention f) Neurological disease other than Parkinson's disease (i.e. multiple sclerosis, stroke) g) Current cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS III | Enrollment On and Off Medications, 6 months post-enrollment, and 12 months post-enrollment
  Rater-observed PD global motor symptoms

SECONDARY OUTCOMES:
Nine Hole Peg Test | Enrollment On and Off Medications, 6 months post-enrollment, and 12 months post-enrollment
  Upper extremity dexterity
Timed Up & Go | Enrollment On and Off Medications, 6 months post-enrollment, and 12 months post-enrollment
  Sit to stand from chair, ambulate 3m, turn, return to chair and sit
Six Minute Walk Test | Enrollment On and Off Medications, 6 months post-enrollment, and 12 months post-enrollment
  Cardiovascular Fitness
Processing Speed | Enrollment On and Off Medications, 6 months post-enrollment, and 12 months post-enrollment
  Symbol/digit matching; test of information processing speed, implicit learning

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No